CLINICAL TRIAL: NCT01480557
Title: Liquefaction Versus Torsional ip. A Comparative Study on Endothelial Cells, Corneal Edema and Corneal Sensitivity
Brief Title: Aqualase Versus Torsional ip. A Study on Endothelial Cells, Corneal Edema and Corneal Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Senior Lecturer, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: liq75tor
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cataract
Keywords: cataract; phacoemulsification; liquefaction; torsional ip; endothelial cell count; central corneal edema; central corneal sensitivity
MeSH Terms: conditions — Cataract | interventions — semen liquefaction factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquefaction group (Active Comparator): Subjects that were operated for cataract using liquefaction technology
  Interventions: Procedure: liquefaction
- Torsional ip group (Active Comparator): Subjects that were operated for cataract using torsional ip technology
  Interventions: Procedure: Torsional ip

INTERVENTIONS:
Procedure: liquefaction — Cataract extraction surgery type
  Arms: Liquefaction group
Procedure: Torsional ip — A type cataract surgery using torsional ip technology
  Arms: Torsional ip group

SUMMARY:
Objective of this study is the comparative assessment of the impact of torsional and liquefaction technologies on endothelial cells (ECC), corneal edema (CCT) and corneal sensitivity (CCS) in a sample of cataract patients.

Participants were recruited from the Cataract Service of the UHA in a consecutive-if-eligible basis. Eligibility criteria included diagnosis of senile cataract with stage 2 nuclear opalescence according to the Lens Opacities Classification System III (LOCS-3) grading scale [10]. By means of a custom computer randomization program all participants randomly populated two study groups according to the cataract-extraction technology used: a) Torsional group (TG) and b) Liquefaction group (LG).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of senile cataract with stage 2 nuclear opalescence according to the Lens Opacities Classification System III (LOCS-3) grading scale

Exclusion Criteria:

* Endothelial cell count less than 1900,
* glaucoma,
* IOP-lowering medications,
* former incisional surgery,
* former diagnosis of corneal disease,
* diabetes or autoimmune diseases

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Endothelial cell count (ECC) | 1 month postoperatively

SECONDARY OUTCOMES:
Uncorrected visual acuity (UVA) | 1 month postoperatively
Central corneal thickness (CCT) | 1 month postoperatively
Central Corneal Sensitivity (CCS) | 1 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Democritus University of Thrace
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Result] Labiris G, Gatzioufas Z, Giarmoukakis A, Sideroudi H, Kozobolis VP. Liquefaction versus torsional IP: a comparative study on endothelial cells, corneal edema and corneal sensitivity. Ophthalmic Res. 2013;49(1):37-42. doi: 10.1159/000342974. Epub 2012 Oct 23. PMID 23095606